CLINICAL TRIAL: NCT04066452
Title: Study of Prevalence of Amyloidosis in Heart Failure (PREVAMIC).
Brief Title: Prevalence of Amyloidosis in Heart Failure (PREVAMIC)
Acronym: PREVAMIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Other Study IDs: FIS-AMI-2019-01
Record Dates: First submitted 2019-08-20; First posted 2019-08-26 (Actual); Last update posted 2020-03-05 (Actual); Status verified 2019-08

CONDITIONS: Heart Failure
Keywords: Amyloidosis
MeSH Terms: conditions — Heart Failure; Amyloidosis | interventions — Urination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single-group studies: Patients will be informed about the study and their written informed consent will be requested.
  Once included in the study:
  * A series of clinical, analytical and echocardiographic parameters will be collected and measured
  * Will be performed:
    * Bone-cardiac scintigraphy with Tc-DPD (or similar: Tc-PYP or Tc-HMDP)
    * Analytical to rule out monoclonal protein:
      * Proteinogram and serum immunoglobulins.
      * Light chains free in serum -Freelite-
      * Immunofixation in serum and urine.
  * The number of readmissions, emergency visits and mortality in the following 12 months will be recorded to compare the readmission and mortality rates in one year of patients with and without CA.
  * The prescribed pre- and post-diagnostic treatments will be described, according to clinical practice (without intervention).
  * No intervention, whether diagnostic or follow-up, that is not the usual clinical practice will be applied to patients.
  Interventions: Diagnostic Test: Bone-cardiac scintigraphy with Tc-DPD (or similar: Tc-PYP or Tc-HMDP).; Diagnostic Test: Proteinogram and serum immunoglobulins. Light chains free in serum -Freelite-. Immunofixation in serum and urine

INTERVENTIONS:
Diagnostic Test: Bone-cardiac scintigraphy with Tc-DPD (or similar: Tc-PYP or Tc-HMDP). — Bone-cardiac scintigraphy with Tc-DPD (or similar: Tc-PYP or Tc-HMDP) to evaluate the degree of cardiac uptake from 0 to 3 degrees.
Diagnostic Test: Proteinogram and serum immunoglobulins. Light chains free in serum -Freelite-. Immunofixation in serum and urine — Analysis to rule out the presence of monoclonal protein in blood and urine.

SUMMARY:
TITLE: Study of Prevalence of Amyloidosis in Heart Failure: PREVAMIC.

DESIGN: Multicenter, observational, cross-sectional, prospective, cohort study with a one-year follow-up. 44 hospitals from Spain will participate.

OBJECTIVES. PRIMARY: To estimate the current prevalence of different types of cardiac amyloidosis (CA) in patients with heart failure, aged 65 years and older, with LVH > 12 mm and any LVEF value, managed in Internal Medicine departments. SECONDARY: To describe the clinical, laboratory and echocardiographic features of patients with CA. To compare one-year readmissions and mortality rates in patients with and without CA.

INCLUSION CRITERIA: Inpatients or outpatients with heart failure, aged ≥ 65 years, both genders, under the care of internists. They should have a NYHA Class II-IV, echocardiogram performed in the previous 24 months, any value of LVEF, LVH: septum or posterior wall > 12 mm, diuretic treatment in the last 6 months and NTproBNP> 1800 pg/ml or BNP> 400 pg/ml in acute hear failure, or NT-proBNP >600 pg/ml o BNP >150 pg/ml in stable condition.

POPULATION: Heart failure outpatients or inpatients of Internal Medicine Services. It is expected to include around 450 patients.

ANALYSIS: To calculate the prevalence of TTR-CA and other types of CA. To compare the clinical, analytical, echocardiographic, and readmissions and mortality rates during one-year in patients with and without CA.

DETAILED DESCRIPTION:
STUDY DESIGN AND PATIENT SELECTION

DESIGN

Multicenter, observational, cross-sectional, prospective, cohort study with a one-year follow-up. Approximately 450 patients will be gathered (according to the calculation of the sample size, 382 patients would be necessary), of both sexes (with stratification Male:Female 1:1), age ≥ 65 years, under the care of Internal Medicine Services, who meet the criteria of the 2016 Heart Failure Guide of the European Society of Cardiology for the diagnosis of Heart Failure, and that have LVH (Septum or Posterior Wall > 12 mm).

Patients will be duly informed of the study and their written informed consent will be requested prior to their enrollment in the study.

Once included in the study a series of clinical, analytical and echocardiographic parameters will be collected and measured.

* It will be performed:

  * Bone-cardiac scintigraphy with Tc-DPD (or similar: Tc-PYP or Tc-HMDP)
  * Analysis to rule out monoclonal protein:

    * Proteinogram and serum immunoglobulins.
    * Free light chains in serum -Freelite-
    * Immunofixation in serum and urine.
* The number of readmissions, emergency visits and mortality in the following 12 months will be recorded to compare the readmission and mortality rates during one year of patients with and without CA
* The prescribed pre- and post-diagnostic treatments will be described, according to clinical practice (without intervention).
* No intervention, whether diagnostic or follow-up, that is not the usual clinical practice will be applied to patients.

POPULATION Inpatients or outpatients of Internal Medicine Services with diagnosis of Heart Failure from the participating centers, selected by the inclusion and exclusion criteria defined for our study, in appropriate number, according to the calculation of the sample size, to assess the main objective.

SELECTION OF HOSPITALS AND PATIENTS All eligible patients will be candidates to enter the study (that is, all those who meet the inclusion criteria and do not meet any exclusion criteria).

The study will involve all Spanish hospitals that voluntarily desire to participate and that have the necessary diagnostic methods to carry out the study. To participate in the study, no minimum hospital size (number of beds) has been set.

DATA COLLECTION AND WORK STRATEGY IN EACH HOSPITAL. The number of cases to be collected by each hospital will be calculated proportionally based on the total number of beds in each center. The number of patients that each center should include refers to the total number of patients.

Data collection will begin the same week of the year for all hospitals. All cases that meet inclusion criteria and none of exclusion and sign the consent will be collected consecutively, with gender stratification (50% men and 50% women of the number of patients assigned to the center) until at least the number of patients assigned to the center is completed . Optionally, patients may continue to be included, in that week or in subsequent weeks,as long as it is done consecutively and stratified by sex (without selecting the cases).

ETHICAL ASPECTS The patients included in this study will be treated according to standard medical care, since being a prevalence study that does not change the usual clinical practice. The study will be carried out in accordance with the Declaration of Helsinki and the Spanish Organic Law on the Protection of Personal Data and Guarantee of Digital Rights.

The study has been approved by the Clinical Research Ethics Committee (CEI) of the Virgen Macarena-Virgen del Rocío University Hospitals. In those cases that are necessary, the approval of the other local CEIs will also be requested.

The researchers of each participating center will explain to each patient all the aspects of the study and the patients will be given an information sheet giving details of it, making it clear that participation is voluntary and that they can leave the study at any time if they wish. If the patient wants to participate, both the investigator and the patient himself, or his legal representative in case of disability, must sign the informed consent. The patient will be given a copy of the consent.

DATABASE An online Database will be developed to record the data of the study patients.

STATISTIC ANALYSIS Continuous variables will be expressed with the value of the mean and standard deviation or as median and interquartile range, depending on the normality of their distribution. Categorical variables will be expressed in percentages or rates. A descriptive analysis of the data will be made, calculating the prevalence rates, and a comparative analysis in relation to different variables, such as gender, age and other factors that are of interest for the objective of the study.

The comparison will be made using the Chi-square test in the categorical variables and the Student's T test for normal quantitative variables. For non-normal quantitative variables, the non-parametric U-Mann Whitney test will be used. Regarding the follow-up data, the association of different variables with the re-entry and mortality data will be assessed using univariate and multivariate analysis. Survival curve analysis will also be performed using the Kaplan-Meier method using log-rank test. A p <0.05 will be considered statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 65 years.
* Both genders
* Heart failure outpatients or inpatients of Internal Medicine Services.
* Heart Failure (Criteria of HF European Guide 2016)
* Symptoms of HF
* NYHA class II to IV
* Echocardiogram performed in the previous 24 months
* FEVI: any value
* HVI: Septum or Posterior Wall > 12 mm
* Diuretic treatment in the last 6 months
* NTproBNP > 1800 or BNP > 400 during any hospital admission, or NTproBNP > 600 or BNP > 150 in a stable situation.

Exclusion Criteria:

* Patients with cancer disease (solid tumor)
* Patients who are included in other studies or clinical trial
* Refusal of patients to participate

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: - Heart failure outpatients or inpatients of Internal Medicine Services of 44 hospitals from Spain. Age ≥ 65 years. Both genders.
Sampling Method: Non-Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2020-02-03 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-09-01 (Estimated)

PRIMARY OUTCOMES:
Prevalence | Through study completion, an average of one year.
  To estimate the current prevalence of different types of Cardiac Amyloidosis in patients with Heart Failure, age ≥ 65 years, with left ventricular hypertrophy (LVH)> 12 mm, and any LVEF value, under the care of internists in different Spanish Hospitals.

SECONDARY OUTCOMES:
Patients characteristics | One year
  To describe the clinical, laboratory and echocardiographic features of patients with CA.
Prognosis | One year
  To compare one-year readmissions and mortality rates in patients with and without AC.

CONTACTS AND LOCATIONS:
Overall Officials: Prado Salamanca Bautista, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (1):
- Hospital Universitario Virgen Macarena, Seville, Spain